CLINICAL TRIAL: NCT02048488
Title: A Phase I/IIa Open-Label, Dose Escalation and Cohort Expansion Trial of Oral TSR-011 in Patients With Advanced Solid Tumors and Lymphomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-20-5006-C
Record Dates: First submitted 2014-01-20; First posted 2014-01-29 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2016-03

CONDITIONS: Solid Tumors; Lymphomas
Keywords: non small cell lung cancer; NSCLC; Anaplastic lymphoma kinase; ALK tyrosine kinase receptor; ALK+; TRK+; ALK inhibitor; TRK inhibitor; tropomyosin receptor kinase; TRKA; TRKB; TRKC; advanced malignancy
MeSH Terms: conditions — Lymphoma; Carcinoma, Non-Small-Cell Lung | interventions — belizatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental Drug TSR-011 (Experimental): Experimental Drug TSR-011
  Interventions: Drug: TSR-011

INTERVENTIONS:
Drug: TSR-011 — Number of cycles until progression or unacceptable toxicity develops.
  Other Names: ALK inhibitor, ALKi; TRK inhibitor

SUMMARY:
TSR-011 is a potent small molecule inhibitor of tyrosine kinases involved in cancer, including:

1. Anaplastic lymphoma kinase (ALK)
2. The tropomyosin-related kinases TRKA, TRKB, and TRKC

This is a sequential, open-label, non-randomized study with dose escalation in Phase 1, followed by expansion at a recommended phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

* To be considered eligible to participate in this study, all of the following requirements must be met:

  1. Patients in Phase 1 must have metastatic or locally advanced solid tumors who have failed to respond to standard therapy
  2. All patients must have confirmation of either ALK positive or TRK positive status.
  3. Patients in Phase 1 will not be required to have measurable disease. All patients in Phase 2a will be required to have measurable disease by RECIST.
  4. All patients enrolled in this study must have tumor tissue available.
  5. Patient (male or female) must be ≥ 18 years of age (except where age of majority is 16 years in a particular country, such as the United Kingdom).
  6. Patient must have performance status ≤2 on the ECOG Performance Scale.
  7. Patient must have an estimated life expectancy of at least 3 months.
  8. Patients must have adequate organ function.
  9. For patients previously treated with myelosuppressive therapy, at least 3 weeks must have elapsed and toxicity must have recovered to grade 1 or baseline. Non-myelosuppressive therapy patients must have recovered from all treatment-related toxicities. Fourteen days must have elapsed since palliative radiation for bone metastasis.
  10. Female patients of childbearing potential must have a negative serum pregnancy test and use adequate birth control for the duration of study participation and for 3 months after the last dose of study drug.
  11. The patient or his or her legal representative must be able to read, understand, and provide signed informed consent.
  12. Patient is able to understand the study procedures and agrees to participate in the study by giving written informed consent.

Exclusion Criteria:

* Patients will not be deemed eligible for entry into this study if any of the following criteria are met:

  1. Patient has leukemia.
  2. Patient is a pregnant or lactating female.
  3. Patient has uncontrolled congestive heart failure, angina, or has had a myocardial infarction in the preceding 3 months.
  4. Ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥2, atrial fibrillation of any grade, or QTc interval >450 msec.
  5. Patients with risk factors for Torsade de point and patients receiving concomitant medication with QT-prolonging medicines.
  6. Patient has an uncontrolled concurrent medical condition or disease.
  7. Patient has undergone bone marrow or stem cell transplantation in the past 6 months.
  8. Patient has a known hypersensitivity to the components of TSR-011 or the excipients.
  9. Patient has active or uncontrolled infection.
  10. Patient has a known psychiatric or substance abuse disorder.
  11. Patient has active second primary malignancy.
  12. Patient is observed to have a clinically active central nervous system (CNS) metastases or carcinomatous meningitis.
  13. Patient has any other severe concurrent disease which, in the judgment of the Investigator, would preclude study participation.
  14. Patient is known to be HIV positive or who has an AIDS-related illness.
  15. Patient has a known history of or active (treated or not) Hepatitis B or C.
  16. Patient has presence of ascites causing significant symptoms.
  17. A patient must stop taking any prescription, over-the-counter, or herbal remedy known to be an inhibitor or inducer of CYP3A4/5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-10; Primary Completion 2016-09 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Approximately 2 years

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC) | Day 1: 0-24 hrs after first dose; pre-dose on days 8 & 15; day 29: 0-24 hours
Maximum Tolerated Dose (MTD) | 28 days after first dose
  Phase 1, during the dose-escalation phase
Response Rate (RR) | approximately 2 years
  Phase 2
Dose limiting toxicity (DLT) | 28 days after first dose
  Phase 1, during the dose escalation phase
Progression Free Survival (PFS) | approximately 2 years
  Phase 2
Recommended Phase 2 Dose (RP2D) | approximately 2 years
  Phase 1

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Bobilev, MD, Study Director — Tesaro, Inc.
Locations (15):
- United States (6):
  - Goodyear, Arizona
  - Scottsdale, Arizona
  - Los Angeles, California
  - Nashville, Tennessee
  - Norfolk, Virginia
  - Spokane, Washington
- Poland (4):
  - Poznan, Greater Poland Voivodeship
  - Warsaw, Masovian Voivodeship
  - Gdansk, Pomeranian Voivodeship
  - Olsztyn, Warmian-Masurian Voivodeship
- Spain (2):
  - Madrid
  - Santiago de Compostela
- Taiwan (2):
  - Tainan
  - Taipei
- London, United Kingdom

REFERENCES:
- [Derived] Lin CC, Arkenau HT, Lu S, Sachdev J, de Castro Carpeno J, Mita M, Dziadziuszko R, Su WC, Bobilev D, Hughes L, Chan J, Zhang ZY, Weiss GJ. A phase 1, open-label, dose-escalation trial of oral TSR-011 in patients with advanced solid tumours and lymphomas. Br J Cancer. 2019 Jul;121(2):131-138. doi: 10.1038/s41416-019-0503-9. Epub 2019 Jun 20. PMID 31217479